CLINICAL TRIAL: NCT06835283
Title: Sequential Accelerated ITBS / Remote tDCS for Treatment of Neuropsychiatric Symptoms in Alzheimer's Disease: A Pilot Study
Brief Title: Novel Brain Stimulation Treatment for Neuropsychiatric Symptoms in Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Ricardo Jorge, MD, Psychiatrist, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-56426
Record Dates: First submitted 2024-12-13; First posted 2025-02-19 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer&Amp;#39;s Disease-related Dementia; Alzheimer Disease; rTMS Stimulation
Keywords: Alzheimer's Disease; tDCS; iTBS; brain stimulation; mood swings
MeSH Terms: conditions — Alzheimer Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: This study investigates a novel approach to managing neuropsychiatric symptoms in Alzheimer's Disease and related dementias using a sequential brain stimulation model. The study combines two techniques: intermittent theta burst stimulation (iTBS) and transcranial direct current stimulation (tDCS). The process begins with in-clinic iTBS sessions to "prime" the brain, potentially enhancing its plasticity and receptiveness to subsequent treatments. This is followed by four weeks of at-home tDCS sessions, administered with caregiver assistance. The sequential use of these treatment methods is based on research suggesting that combining techniques may amplify therapeutic effects. The study aims to evaluate both the feasibility of this approach and its potential effects on symptoms and brain function, providing insights for future larger clinical trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Brain Stimulation (Other): Participants will receive a combination of two non-invasive brain stimulation treatments. During the first week, iTBS sessions will be administered in-clinic for five consecutive days, using magnetic pulses to target brain areas associated with neuropsychiatric symptoms. This is followed by four weeks of daily, self-administered tDCS at home, delivering a low electrical current to modulate brain activity. Participants will complete brain scans and questionnaires at various points to evaluate changes in the brain and symptom severity.
  Interventions: Device: Brain Stimulation

INTERVENTIONS:
Device: Brain Stimulation — This intervention is distinct because it combines two non-invasive brain stimulation techniques, intermittent theta burst stimulation (iTBS) and transcranial direct current stimulation (tDCS), in a sequential manner. Unlike studies that evaluate these techniques individually, this study explores their combined and complementary effects, with iTBS priming the brain to enhance the subsequent impact of tDCS. The sequential design leverages different mechanisms of action: iTBS delivers magnetic pulses to targeted brain areas to modulate neural activity, while tDCS applies a low electrical current for sustained modulation. This approach specifically targets neuropsychiatric symptoms (e.g., mood swings, apathy, and agitation) in individuals with Alzheimer's Disease and related dementias (ADRD), a population often underserved by traditional interventions. The study also evaluates the feasibility of at-home tDCS administration, making it unique in combining clinical and caregiver-managed treat

SUMMARY:
The goal of this pilot study is to test a combination of two non-invasive brain stimulation methods, called iTBS (intermittent theta burst stimulation) and tDCS (transcranial direct current stimulation), in people with Alzheimer's Disease (AD) and related dementias (ADRD). This study will also explore whether the combined treatment shows promise for reducing neuropsychiatric symptoms like mood swings, apathy, and agitation, and will evaluate the impact of the treatment on caregivers.

The main questions the study aims to answer are:

1. Is the combined brain stimulation treatment practical and well-tolerated?
2. Do preliminary results suggest that this treatment could help manage neuropsychiatric symptoms and support a larger study?

Participants will:

* Attend nine in-person visits over three months.
* Complete one week of in-clinic brain stimulation sessions (iTBS) followed by four weeks of daily at-home brain stimulation sessions (tDCS).
* Take part in brain scans, questionnaires, and brain activity tests before and after the treatment.

This pilot study is a first step to assess whether this combined treatment approach is practical and whether it has potential to improve symptoms, laying the groundwork for larger studies in the future.

DETAILED DESCRIPTION:
This study is designed to explore a new way to manage behavioral and emotional symptoms in people with Alzheimer's Disease (AD) and related dementias (ADRD). Many people with these conditions experience mood swings, apathy, or agitation, which can be difficult to treat with current medications due to limited effectiveness and side effects. This research is testing whether two types of brain stimulation, called iTBS (intermittent theta burst stimulation) and tDCS (transcranial direct current stimulation), can be combined to provide a non-invasive and potentially effective treatment for these symptoms.

Brain stimulation is already used in other areas of medicine and involves applying gentle magnetic or electrical stimulation to the brain. iTBS uses short bursts of magnetic pulses, while tDCS uses a low electrical current. Both methods are painless, safe, and do not require surgery. This study is the first to look at combining these two techniques for people with AD/ADRD, based on findings from other research that suggest the combination might have stronger effects than either method alone.

Since this is a pilot study, the focus is on understanding whether the treatment process is practical for both patients and caregivers. This includes evaluating how easy it is for participants to attend the clinic sessions, whether caregivers can successfully administer the at-home treatments, and whether the overall process is manageable for families. In addition to these practical questions, researchers will also collect preliminary data to see if the treatment helps improve behavioral symptoms and measure any changes in the brain using scans and brain activity tests.

Participants will spend one week receiving treatments in a clinic and four weeks using a portable device for at-home sessions. Researchers will closely monitor participants throughout the study to ensure safety and will follow up to see if any improvements last after the treatment ends.

The study is an important step in understanding whether this new approach has potential to help people with AD/ADRD and whether it should be studied further in larger trials. It also aims to identify how to make the treatment process as smooth and effective as possible for patients and caregivers.

ELIGIBILITY:
Inclusion criteria

1. veteran between the ages of 60 to 85
2. clinical diagnosis of mild to moderate Alzheimer's disease or related dementia
3. clinically significant neuropsychiatric symptoms (NPS) evidenced by a score ≥ 2 in at least one domain of the Neuropsychiatric Inventory Questionnaire
4. mild to moderate cognitive impairment demonstrated by a Mini-Mental State Examination (MMSE) score of 15-23
5. have a caregiver who is able and willing to escort the patient to/from clinic visits, answer questionnaires, and assist in the implementation of treatment sessions at home
6. if taking psychotropic medications, demonstrate stability for at least 4 weeks of treatment

Exclusion Criteria:

1. any contraindication for MRI
2. any contraindication for iTBS/tDCS including but not limited to seizure disorder, severe cardiovascular disease, history of brain surgery, or stroke involving the cerebral cortex near area of stimulation
3. current alcohol or substance use disorder determined by QuickSCID (nicotine allowed; mild cannabis and alcohol use is allowed)
4. neuropsychiatric symptoms (NPS) that are severe enough to preclude the intervention from being delivered safely and effectively, particularly agitation or aggression.

6) any unstable coexisting medical condition that in the opinion of the principal investigator(s) interferes with the treatment protocol or increase the likelihood of adverse events.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of iTBS-tDCS treatment in ADRD patients | From enrollment until the end of treatment at 5 weeks
  The feasibility of providing sequential iTBS-tDCS treatment to ADRD patients with neuropsychiatric symptoms is a primary focus. Feasibility will be assessed mainly through rates of by recruitment, retention and adherence. Recruitment rate is the number of enrolled patients divided by the total number of patients who initially approached the study or had interest in it. Retention rate is the percentage of patients who complete the entire study out of the initial enrolled participants, and then adherence rate is the number of completed iTBS and tDCS sessions divided by the total prescribed treatment sessions. Since feasibility is being evaluated as the primary aim instead of efficacy, there is no randomization or probability of group assignment. Each and every subject will undergo the same treatment stimulation process, as they will all have 1 week of in-clinic iTBS sessions and then four weeks of at-home tDCS sessions.
Tolerability of iTBS-tDCS treatment in ADRD patients | From enrollment until the end of treatment at 5 weeks
  The tolerability of providing sequential iTBS-tDCS treatment to ADRD patients with neuropsychiatric symptoms. Tolerability will be evaluated based on the frequency and severity of adverse events reported during the intervention period. These findings will inform the design and implementation of a larger clinical trial.

SECONDARY OUTCOMES:
Neuropsychiatric Symptoms | From enrollment until the end of treatment at 5 weeks
  We will gather preliminary data on the potential effects of iTBS-tDCS on neuropsychiatric symptoms in individuals with Alzheimer's Disease and related dementias, as determined by changes in standardized neuropsychiatric symptom questionnaires pre- and post-treatment.
Caregiver burden | At baseline (week 0) and post-treatment (week 6)
  We will also explore the potential impact of the treatment on caregiver burden using caregiver-reported outcomes collected before and after the intervention. The total score of caregiver burden will involve the sum of the responses to all items on the Zarit Burden Interview assessment, and these scores are rated on a Likert scale of 0-4. This total score quantifies the level of caregiver burden, as high scores will indicate greater burden. Descriptive statistics; such as mean, median, and standard deviation-will summarize the overall caregiver burden within the study sample. Other factors associated with determining caregiver burden include inferential statistical methods like multiple regression analysis or ANOVA, as these will be used to examine connections between ZBI scores and variables such as patient cognitive function, treatment compliance, and demographic factors.
Brain connectivity through MRI | At baseline visit (week 0) and post-treatment (week 6)
  We can observe potential changes in brain connectivity through functional MRI scans conducted pre- and post-treatment, to inform hypotheses for future studies. The MRI will be used to obtain baseline images and neuromodulation-induced changes of brain structure as well as functional connectivity, particularly in the default mode and salience networks.

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

REFERENCES:
- [Background] Ahn H, Sorkpor S, Miao H, Zhong C, Jorge R, Park L, Abdi S, Cho RY. Home-based self-administered transcranial direct current stimulation in older adults with knee osteoarthritis pain: An open-label study. J Clin Neurosci. 2019 Aug;66:61-65. doi: 10.1016/j.jocn.2019.05.023. Epub 2019 May 29. PMID 31153751